CLINICAL TRIAL: NCT04718558
Title: Evaluation of the Effect of Boyle-Davis Mouth Gape on Intracranial Pressure in Patients With Cleft Palate Repair by Measuring Optic Nerve Sheath Diameter
Brief Title: Optic Nerve Sheath Diameter Measurement in Cleft Palate Repair
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, assistant professor, Karadeniz Technical University
Other Study IDs: 2020/271
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Cleft Palate
Keywords: optic nerve sheat diameter; mouth gag; cleft palate; ultrasonography
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged between 3-24 month and undergoing cleft palate surgery

SUMMARY:
The aim of this study is to evaluate the effect of the Boyle-Davis mouth opener, which is routinely used in cleft palate surgery, on intracranial pressure by USG-guided optic nerve sheath diameter measurement, which is a non-invasive method with proven effectiveness and reliability in recent years.

DETAILED DESCRIPTION:
Non-syndromic cleft lip and / or palate is a complex congenital defect that results from multiple genetic and environmental factors. It is also one of the most common congenital malformations. Cleft defects require early surgical repair to minimize nutritional difficulties and ensure optimum speech function. The Boyle-Davis mouth opener used in cleft palate surgery consists of tongue blade, mouth opener and suspension system and is used to fix the endotracheal tube in the midline and provide excellent surgical vision during the operation. However, it can cause complications such as dental injuries, laryngospasm, and displacement of the tracheal tube.

Undesirable effects such as changes in heart rate and increases in intracranial pressures may occur during endotracheal intubation. These hemodynamic responses are thought to be due to increased sympathoadrenal activity. Laryngoscopy without tracheal intubation has been shown to increase high catecholamine levels and blood pressure, suggesting that sympathoadrenergic response occurs more frequently due to stimulation of the supraglottic region. Although the Boyle-Davis mouth opener provides an advantage for access to the intraoral cavity, its insertion causes significant increases in intracranial pressure (ICP) and intraocular pressures by causing hemodynamic changes similar to laryngoscopy.

In recent studies, measurement of optic nerve sheath diameter with ultrasonography, which is a non-invasive method, is frequently used in the detection of intracranial pressure increases. The optic nerve is a part of the central nervous system and is covered with a dural sheath. Pressure changes in the intracranial region are similar to the pressure in the infraorbital subarachnoid space surrounding the optic nerve. In clinical studies, it has been shown that changes in intracranial pressure correlate with the optic nerve sheath diameter measured by ultrasonography. Compared to other diagnostic methods, measurement of the diameter of the optic nerve sheath is an inexpensive, easy-to-apply and non-invasive method. In our study, we aimed to determine the intracranial pressure changes that may occur due to the use of mouth gag in cleft palate surgeries by measuring the optic nerve sheath diameter with USG, which is a non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 3-24 month and with an ASA physical status I-II and undergoing cleft palate surgery will be included to the study.

Exclusion Criteria:

* Exclusion criteria will be preexisting acute or chronic eye disease,
* History of eye surgery, use of drugs known to influence intraocular pressure (IOP) (ß blockers, Ca channel blockers, statins and nitrates)
* Conditions that may cause known intracranial pressure changes (cerebrovascular event, bleeding, an intracranial tumor, etc.)
* patients' parental refusal

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged between 3-24 month and with an ASA physical status I-II and undergoing cleft palate surgery will be included to the study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
change in optic nerve sheath diameter | After general anesthesia induction, after endotracheal intubation, after mouth gag insertion (primary timepoint), 20 minutes, 40 minutes, 60 minutes after mouth gag insertion
  Change in optic nerve sheath diameter as assessed by rapid ultrasound scan before general anesthesia, after intubation, 1 minute, 10 minutes, 20 minutes, 40 minutes, 60 minutes after mouth gag is inserted and after mouth gape is removed

SECONDARY OUTCOMES:
Change in heart rate | After general anesthesia induction, after endotracheal intubation, after mouth gag insertion (primary timepoint), 20 minutes, 40 minutes, 60 minutes after mouth gag insertion
  Change in heart rate by using electrocardiogram on the anesthesia workstation
Change in End tidal CO2 | After general anesthesia induction, after endotracheal intubation, after mouth gag insertion (primary timepoint), 20 minutes, 40 minutes, 60 minutes after mouth gag insertion
  Change in End tidal CO2 by using capnography on the anesthesia workstation
Change in Peak inspiratory pressure (PIP) workstation | After general anesthesia induction, after endotracheal intubation, after mouth gag insertion (primary timepoint), 20 minutes, 40 minutes, 60 minutes after mouth gag insertion
  Change in Peak inspiratory pressure (PIP) by using monitoring on the anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)